CLINICAL TRIAL: NCT05662501
Title: Non Randomised, Prospective, Single Center Clinical Study to Evaluate the Safety and Procedural Feasibility of an Innovative Flow Assist Device, Pleioflow-RF.
Brief Title: Pleiades Safety and Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pleioflow (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PLEIO21
Record Dates: First submitted 2022-06-18; First posted 2022-12-22 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Elective Cardiac Surgery
Keywords: acute kidney injury; cardiac surgery; flow assist; intra-aortic balloon pump; renal failure
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects receiving the Pleioflow-RF device (Experimental): Subjects receiving the Pleioflow-RF device in conjunction with IABP
  Interventions: Device: Pleioflow-RF

INTERVENTIONS:
Device: Pleioflow-RF — Subjects who are going to undergo scheduled cardiac surgery and are prone to developing renal insufficiency, will receive the Pleioflow-RF device in conjunction with IABP during CPB. Subjects will be followed until 30-days post-intervention.

SUMMARY:
The "Pleiades" study is a non randomised, prospective, single center clinical trial that aims to evaluate the safety and the procedural feasibility of an innovative flow assist device (Pleioflow-RF) in adult patients undergoing elective cardiac surgery.

DETAILED DESCRIPTION:
This is a non randomised, prospective, single center clinical study that aims to evaluate the safety and the procedural feasibility of an innovative flow assist device (Pleioflow-RF) in adult patients, undergoing elective cardiac surgery. The Pleioflow-RF is a percutaneous flow assist device that functions in combination with the traditional Intra Aortic Balloon (IAB). It represents a modified, probably improved, safer and more potent version of the latter, with respect to its dramatic ability to increase renal perfusion in low flow and pressure conditions -as displayed in large animal trials.

The Pleioflow RF -IAB assembly integrates two critical elements:

(i) a soft Nitinol stent element, positioned at the tip of the IAB, deployed in the descending Aorta that centralizes the IAB, thus preventing excessive IAB movement, protecting the wall of the Aorta from IAB induced injury, and the renal arteries from occlusion, (ii) a downstream valve, mounted within the above stent, that keeps the pressure and flow augmentation, created by the IAB's periodic inflation, localised below said valve, in the abdominal Aorta, where the renal arteries originate.

The device is used intraoepratively, during Cardiopulmonary by pass (CPB). During IAB inflation, the IAB occupies space and the pressure increases instantly. The downstream valve above the IAB, receives this pressure wave and closes. The valve closure blocks upstream flow, and diverts all the flow and pressure wave generated by the IAB primarily towards the kidneys and the periphery.

Due to the continuous IAB's perdiodic inflation and deflation, the device converts the constant CPB flow and pressure to pulsatile, towards the kidneys.

The device is expected to increase substantially the renal perfusion during Cardiac Surgery; it may therefore decrease the post-operative incidence of renal failure.

The hypothesis of this clinical study is that the placement of the Pleioflow-RF intraoperatively, particularly in patients who are more prone to developing renal deterioration based on either their Cleveland Clinic prognostic score, or/and the pre-existence of renal impairment, can prevent further renal deterioration in these patients. These vulnerable patients comprise 10-20% of the total cardiac surgery population.

Following informed consent, subjects eligible for a elective cardiac surgery that meet all of the inclusion, and none of the exclusion, criteria will be enrolled into the study. The Pleioflow-RF will be inserted preferrably through a 9F sheath into the femoral artery; then advanced into the descending thoracic aorta, and positioned below the origin of the left subclavian artery under transoesophageal echocardiography guidance. Subsequently through the same sheath, the intra-aortic balloon (IAB) will be placed and be advanced up to the proximal tip end of the Pleioflow-RF device. The IABP will be connected to an IAB pump. The duration of operation of the assembly (Pleioflow-RF and the IAB) will be for as long as the cardiopulmonary bypass(CPB) time, in order to protect the kidneys from hypoperfusion, during that time. After the end of the CPB, the IABP and the device will be removed. Subjects will be followed up until 30 days post intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 85, men and women
2. Elective coronary artery bypass grafting surgery and/or heart valve surgery with planned CPB.
3. Written informed consent provided
4. Haemoglobulin (Hb) ≥ 11 g/dl in women and ≥ 12 g/dl for men
5. Ejection fraction ≥ 30%
6. Score≥ 3 according to the Cleveland Clinic Foundation risk factor scale for AKI and / or Chronic Kidney Disease (CKD) with preoperative glomerular filtration rate, estimated glomerular filtration rate, eGFR ≤50 ml / min / 1.7, 3 m2) as estimated by the equation of four Modified Diet and Renal Disease variables (MDRD type)

Exclusion Criteria:

1. emergency surgery
2. severe sepsis or rhabdomyolysis
3. severe preoperative renal insufficiency requiring renal replacement therapy (RRT) or even once RRT
4. receiving within the last 10 days nephrotoxic medications, such as radiocontrast material (> 100 ml), amphotericin B, aminoglycosides, NSAID, or trimethoprim-sulfamethoxazole with at least moderate renal impairment (eGFR ≤45)
5. Any severe coagulopathy
6. Participation in another trial
7. Any surgical or medical condition which according to investigator's opinion could create problem in the assessment of safety and /or efficacy of the device
8. Severe comorbidity with life expectancy < 6 months
9. History of poor compliance with previous treatment and incapability of giving informed consent
10. Pregnant or breastfeeding women. Pregnancy, confirmed by a positive laboratory test for Human Chorionic Gonadotropin, is considered from the time after conception until the end of the pregnancy.
11. Peripheral artery disease making insertion of IABP unfeasible
12. Preoperative intra-aortic balloon pump (IABP)
13. Preoperative other device in the same anatomical area (which could possibly create dysfunction of any of the other two devices)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Pleioflow-RF device | Through end of Device removal procedure
  Feasibility: Initiation and maintenance the Mean of the maxima (maximum values) of pulsatile pressure ≥65mmHg during cardiopulmonary bypass (CPB)
Safety of the Pleioflow-RF device | Through end of Device removal procedure
  Safety: Major Device-Related Adverse Events

SECONDARY OUTCOMES:
Duration of Intensive Care Unit/Intensive Therapy Unit (ICU/ITU) stay | 30 days
Duration of Hospital Stay | Up to 30 days postoperative
Acute Kidney injury (AKI) | Up to 7 days postopoerative
Need for renal replacement therapy | Up to 7 days
Intraoperative and Postoperative use of inotropes and vasopressors | Up to 7 days postoperative
  Number of days and dose of inotropes and vasopressors
30-Day All-Cause Mortality | 30 days
Device- related adverse events | 30 days
Evaluation of clinical data. | Up to 4 hours
  Recording the haemodynamic data: arterial pressure above and below the device
Levels of biomarkers. | Up to 7 days
  Recording the following biomarkers levels: Creatinine, Urea, electrolytes and Neutrophil gelatinase associated lipocalin (NGAL)
Conversion of non- pulsatile to pulsatile flow and pressure during CPB | Up to 4 hours
Mean of Maximum pulsatile pressure values peripherally to the valve of the Pleiofow-RF device | Up to 4 hours
  Mean of Maximum pulsatile pressure values peripherally to the valve of the Pleiofow-RF device, greater than or equal to 80 mmHg (≥ 80 mm Hg), or increase of Mean of maxima (maximum values of pulsatile pressure), peripherally to the valve of the Pleiofow-RF device≥ 20 mmHg above the mean arterial pressure (MAP) of the non pulsatile flow of the extracorporeal circulation, the latter being recorded 2 minutes prior to the activation of the device
Incidence of Pleioflow-RF Device's dysfunction and failures | Through end of Device removal procedure
Measure of ease of device insertion delivery, deployment, positioning | At time of device insertion
  Each assessment (insertion, delivery, deployment, and positioning) will be measured independently using the same unit according to the Procedure feasibility score scale as described in the Appendix 1 in the Protocol. A scale (Procedure feasibility score scale as described in the Appendix 1 in the Protocol) will be used to assess the aforementioned outcome. Minimum value is 1 and maximum value is 5, with higher scores stating a better outcome.
Measure of ease of device removal | Through end of Device removal procedure
  A scale (Procedure feasibility score scale as described in Appendix 1 in the Protocol) will be used to assess the aforementioned outcome. Minimum value is 1 and maximum value is 5, with higher scores stating a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Stavridis, Principal Investigator — Onassis Cardiac Center
Locations (1):
- Onassis Cardiac Center, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided